CLINICAL TRIAL: NCT05973214
Title: Effectiveness of a Cognitive and Behavioral Treatment Program in People With Idiopathic Environmental Intolerance (IEI)
Acronym: BELIEFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C22-19; 2022-A01370-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Environmental Intolerance
Keywords: Environmental health; Idiopathic Environmental Intolerance; Cognitive Behavioral Therapy; Functional Disorder; Somatic Symptoms
MeSH Terms: conditions — Multiple Chemical Sensitivity; Medically Unexplained Symptoms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Parallel two-armed randomized controlled study with a waitlist control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Waitlist (Other)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT for IEI

SUMMARY:
Idiopathic Environmental Intolerance (IEI) denotes a functional disorder represented by heterogeneous symptoms that sufferers attribute to specific environmental agents and for which there may be no solid evidence of an underlying physiological cause.

We are conducting a randomized controlled trial study to compare patients before and after a newly developed cognitive behavioral therapy treatment program for IEI, with respect to behavioral and psychometric variables.

The results of this research project are expected to contribute to advancements in the clinical treatment of IEI, as well as to elaborate on existing theoretical models of IEI.

DETAILED DESCRIPTION:
Introduction:

A percentage of the population report various, nonspecific somatic and cognitive symptoms (e.g., headaches, nausea, fatigue, difficulty concentrating...) that they causally attribute to agents in their environments (chemicals, electromagnetic fields, windmills..). This condition is called Idiopathic Environmental Intolerance (IEI). It is proposed that the attribution of symptoms to an environmental agent, and the associated negative expectations is what drives symptom experience. We hypothesize that this, alongside other cognitive biases, are involved in the emergence and maintenance of symptoms. Treatment models have been developed, but no cognitive behavioral therapy was tested on IEI patients.

The planned study aims to investigate the feasibility and efficacy of a cognitive behavioral treatment online program, in ameliorating quality of life in a French population of patients suffering from IEI.

Methods and analysis:

This parallel two-armed, randomized controlled trial, evaluates an 8-week guided intervention against a wait-list control group. It is a hybrid intervention that will include web-based consecutive modules based on disorder-specific cognitive behavioral therapy (CBT) as well as general transdiagnostic principles . Guidance will be provided by trained psychologists with weekly supportive feedback.

As part of the "BELIEF" project, the present study aims to recruit n=82 patients indicating symptom attributed to factors in the environment. Assessments will take place at baseline and after intervention completion (12 and 24 weeks after randomization). The primary outcome will be measured by the SF-12 scale for quality of life. Secondary outcomes include symptom perception, severity and distress, eco-anxiety, emotional processing, intolerance to uncertainty and associated mental disorders such as depression and anxiety. Consumption of healthcare services will also be measured.

Ethics and dissemination:

Ethics approval has been granted. Results from this study will be published in peer-reviewed journals and presented at international conferences.

Trial registration number: DRKS00014375

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years,
* Present a diagnosis of idiopathic environmental intolerance confirmed by the lead physician at the admission
* Be affiliated to a social security regime.
* Informed Consent

Exclusion Criteria:

* Severe depression, delusion disorder or substance use disorder
* No access to internet
* Non-French speakers
* Currently participating to another research on IEI
* Under an exclusion period for another study
* Benefiting from French state aid known as AME
* Deprivation of liberty by court or administrative order
* Hospitalized without consent
* Under protective measures
* Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey - 12 | T0; 3 Months ; 6 Months
  Measures quality of life with a minimum value of zero and a maximum value of 100. Higher score indicates better outcome.

SECONDARY OUTCOMES:
The Somatic Symptom Disorder - B Criteria Scale | T0; 3 Months ; 6 Months
  Measures criteria for Somatic Symptom Disorder (SSD) and symptoms' burden: The total score ranges between 0 and 48, with a higher score reflecting higher levels of the psychological features of the SSD, or worse outcome.
Symptom Interpretation Questionnaire | T0; 3 Months ; 6 Months
  Measures causal attributions individuals make of common somatic symptoms by using three sub scales: somatic (range 13-36), psychological (range: 13-52), and environmental/normalizing (range: 17-49). Each sub score represents the extent with which each sub scale is endorsed as a possible cause for symptoms (higher score means higher outcome).
QEESI (Quick environnemental exposure and sensitivity inventory) | T0; 3 Months ; 6 Months
  Measures Chemical Sensitivity with 5 subscales: Symptoms, Chemical Intolerances, Other Intolerances, Masking, and Life Impact.
  Patients with no intolerance to chemicals only complete the subscales on Symptoms.
11-item Electromagnetic Field Sensitivity Scale | T0; 3 Months ; 6 Months
  Measures sensitivity to Electromagnetic Fields. The score can range from 0 to 54 (high score representing high annoyance/intolerance and worse outcome). Only patients reporting intolerance to Electromagnetic fields complete this questionnaire.
Modern Health Worries Scale short (12-item) version | T0; 3 Months ; 6 Months
  Measures Modern Health Worries (concerns of respondents about modern environmental issues). Scores range from 12 to 60 with higher scores indicating more concern or worse outcome.
Climate Change Anxiety Scale | T0; 3 Months ; 6 Months
  Measures Climate Change Anxiety with scores ranging from 13 to 65 and higher scores indicating higher levels of climate change anxiety, or worse outcome.
Hospital Anxiety and Depression scale | T0; 3 Months ; 6 Months
  Measures Depression and Anxiety. Score ranges from 0 to 21 with higher score representing worse outcome.
Short version of the Intolerance of Uncertainty Scale | T0; 3 Months ; 6 Months
  Measures Intolerance to Uncertainty with total scores ranging from 12 to 60 with higher score representing worse outcome. The total scores encompasses two sub-scales: prospective anxiety and inhibitory anxiety. A greater score in each subscale indicates a greater level of prospective anxiety and inhibitory anxiety.
Body Perception Questionnaire - Very Short Form | T0; 3 Months ; 6 Months
  Measures body awareness and autonomic stress response patterns. Scores range from 12 to 60. Particularly high scores may indicate the autonomic nervous system is frequently activated by stress or chronic threat responses (i.e. worse outcome)
Levels of Emotional Awareness Scale 10 item | T0; 3 Months ; 6 Months
  Measures the Level of Emotional Awareness with a maximum score of 50. Higher scores indicating greater awareness and differentiation in emotions, or better outcome.

OTHER OUTCOMES:
Attitudes Towards Seeking Mental Health Services Inventory (IASMHS) | T0
  measures how people think and feel regarding utilizing psychological healthcare. This 24-item scale assesses 3 internally consistent factors: psychological openness, help-seeking propensity, and indifference to stigma. Participants answer the questions using a 5-item scale (0 = disagree; 4= agree). Higher scores on the indifference to stigma scale reflect a positive stance towards mental healthcare services, while higher scores on the other two subscales reflect a more negative attitude.
healthcare utilization questionnaire | T0, 3 months, 6 months
  Consists of 6 questions with an open answer format and assesses the number of medical and paramedical visits, therapists' visits, physical exams, as well as medication and dietary supplements consumed over the last 3 months.
Working Alliance Inventory | filled out after 3 weeks into treatment by the therapist.
  Measure three dimensions of working alliance: agreement on therapeutic goals, consensus on tasks, and affective bond between client and therapist. The questionnaire consists of eight items measured on a five-point scale (1=never to 5=always), as well two open questions for feedback to the therapist. A higher score indicates a better client-therapist relationship.
Affect and Symptom Paradigm | t0, 3 months, 6 months
  Studies how negative affective stimuli influence somatic symptom perception. Negative and neutral pictures are presented to participants and after each picture series, participants fill in a short questionnaire about their current symptoms and affective state.
Attribution Bias task | t0, 3 months, 6 months.
  Monitors symptoms during 2X10 mins exposure to environmental agents patients attribute symptoms to (wifi box or chemicals) and 1X10 mins control without exposure. Patients can stop the task at all times.
Belief Updating Task | t0, 3 months, 6 months.
  This task was developed to investigate information processing and belief updating in light of desirable or undesirable information. Patients rate their own risk for negative events, some of them related to environmental hazards, as compared to baseline risks in the general population.
Client Satisfaction Questionnaire | either 3 months (intervention group) or 6 months (waitlist group)
  Explores patients' feedback after receiving the traitement protocole, in 8 questions from 1 to 4 (high score representing high satisfaction) and 2 open questions for comments and suggestions.

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Lemogne, PR, MD, Principal Investigator — Institut de Psychiatrie et des Neurosciences de Paris
Locations (1):
- Unité de pathologies professionnelles et environnementales, Hôtel-Dieu, Paris, Paris, France